CLINICAL TRIAL: NCT06384950
Title: Evaluating the Role of ChatGPT in Educating Patients With Early-stage Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2023-11-005A
Record Dates: First submitted 2024-04-16; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Carcinoma, Hepatocellular
Keywords: ChatGPT; Patient Education
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: To compare the educational effectiveness of a chatbot integrated with health education information to traditional health education methods. This comparison encompassed aspects such as the patient's health literacy and clinical satisfaction. Based on the findings, recommendations and improvements would be proposed to promote the application and development of large language models in the medical field.
Who Masked: Participant
Masking Description: The research uses a Randomized Controlled Trial (RCT) methodology, dividing patients into a control group undergoing the conventional patient education routine, and an experimental group that leverages both the chatbot and traditional education. By comparing selected outcomes between the two groups, the experiment's effectiveness will be determined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPT-3.5-based educational (Experimental): Patients receive additional education using a GPT-3.5-based educational robot on top of the traditional education.
  Interventions: Behavioral: ChatGPT
- Traditional education procedures (Active Comparator): Patients receive standard traditional education procedures.
  Interventions: Behavioral: patient education with traditional methods.

INTERVENTIONS:
Behavioral: ChatGPT — Patients receive additional education using a GPT-3.5-based educational robot on top of the traditional education.
  Other Names: Add GPT-3.5 model for patient education
  Arms: GPT-3.5-based educational
Behavioral: patient education with traditional methods. — Patients receive standard traditional education procedures.
  Arms: Traditional education procedures

SUMMARY:
Liver cancer is a leading cause of cancer-related deaths in Taiwan, with its onset linked to factors like chronic liver conditions, cirrhosis, and genetic predispositions. According to the "Barcelona Clinic Liver Cancer (BCLC)" classification, early-stage liver cancer is demarcated by stages 0 to A. Upon such diagnosis, both patients and their families often have numerous questions and concerns, ranging from treatment choices to long-term outcomes. The research proposes a GPT-3.5-based chatbot to assist these patients by providing timely, personalized information, aiming to enrich their understanding of the disease and improve communication between patients and health professionals.

The research methodology employs a Randomized Controlled Trial (RCT) design, dividing participants into a control cohort receiving standard patient education routine and an experimental cohort receiving both the AI chatbot and traditional education routine. The comparative analysis of these cohorts will determine the effectiveness of the AI intervention in improving patients' health literacy and satisfaction.

DETAILED DESCRIPTION:
Liver cancer is the second most common cause of cancer-related deaths in Taiwan. Various factors play a role in its development, such as chronic liver conditions, cirrhosis, viral infections, alcohol intake, obesity, diabetes, and genetic predispositions, among others. Based on the "Barcelona Clinic Liver Cancer (BCLC)" system, early-stage liver cancer falls within stages 0 to A. When faced with an early-stage liver cancer diagnosis, patients and their relatives frequently express concerns. These may range from the potential effects of the disease on daily living, evaluating treatment options, potential side effects, costs involved, the chances of recurrence, and survival rates, to the care required after the treatment. Addressing these worries often requires extensive explanations and time for the patients to process the information.

The research proposes using a chatbot built upon the GPT-3.5 language model developed by OpenAI for patient education services. Such a chatbot would aid early-stage liver cancer patients navigate the complexities of obtaining relevant information. As an artificial intelligence technology, the chatbot can offer timely, personalized information and psychological support. By responding to patients' inquiries, the chatbot can provide a thorough understanding of basic liver cancer knowledge, its causes, and treatment approaches, thereby facilitating a deeper comprehension of the early stages of liver cancer and its treatment regimen. Patients and their relatives can comprehend their condition and treatment plans, enhancing their conversations with medical staff and promoting a harmonious doctor-patient relationship.

The research uses a Randomized Controlled Trial (RCT) methodology, dividing patients into a control group undergoing the conventional patient education routine, and an experimental group that leverages both the chatbot and traditional education. By comparing selected outcomes between the two groups, the experiment's effectiveness will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early-stage hepatocellular carcinoma from both gastroenterology and general surgery outpatient departments were included. Early-stage hepatocellular carcinoma is defined based on the Barcelona Clinic Liver Cancer (BCLC) staging as stages 0 to A.

Exclusion Criteria:

* Patients under the age of 18 or those currently undergoing treatment for other cancers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-11-29 (Estimated); Study Completion 2025-03-21 (Estimated)

PRIMARY OUTCOMES:
Health literacy score of patients | 1 weeks to 1 month
  Primarily measured using the Liver Cancer Knowledge Scale. The scale consists of 20 questions with options including correct, incorrect, and unsure, with 14 correct answers and 6 incorrect ones (questions 4, 7, 11, 15, 18, 19). Each correct answer scores 5 points, while incorrect or unsure answers score 0 points. The score range is from 0 to 100, with a total score of 100 points.
Satisfaction score with medical care | 1 weeks to 1 month
  It mainly includes satisfaction with traditional health education and AI-based health education tools. The Likert scale assessed the score, which offers options ranging from very dissatisfied (1) to very satisfied (5).

SECONDARY OUTCOMES:
Degree of patient anxiety | 1 weeks to 1 month
  Measured using The GAD-7 questionnaire, a scale designed to assess anxiety levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: No